CLINICAL TRIAL: NCT01816386
Title: Acupuncture Randomized Trial for Post Anaesthetic Recovery and Postoperative Pain - a Pilot Study
Brief Title: Acupuncture Trial for Post Anaesthetic Recovery and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Johannes Fleckenstein, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AcuARP
Record Dates: First submitted 2012-10-28; First posted 2013-03-22 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Laparoscopic Surgery of Uterus, Adnex or Ovaries; Postoperative Pain
Keywords: acupuncture; anaesthetic recovery; perioperative care; Age 18+; ASA-score ≤ 2; Surgery: Uterus; Surgery: Adnex; Surgery: Ovaries
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture Regimen (Active Comparator): Standard anaesthetic procedure plus press needle acupuncture
  Interventions: Other: Acupuncture Regimen
- Standard Treatment Control (No Intervention): Standard anaesthetic procedure plus No treatment.
  All standardized medication according to the perioperative anaesthetic guideline, Department of Anaesthesiology, University of Munich, will be allowed. In special:
  According to the guidelines, anxiolysis will be performed intravenously according to the standard guidelines with opioid immediately prior to the induction of anaesthesia.
  Intraoperative anaesthesia will be performed according to our in-house guidelines: on general recommendations and guidelines of the German society for anaesthesiology (DGAI). Opioids and propofol will be administered via TCI pumps according to the standard protocol.
  It is allowed to treat the subject for pain with metamizol (4*1.25 g/day) and additional piritramide (PCA; 2 mg each 10 minutes; maximum dosage 30 mg/4 hours) .
  Variation of this guideline based regimen are allowed if medically indicated.
- Acupressure Regimen (Active Comparator): Standard anaesthetic procedure plus press plaster acupressure
  Interventions: Other: Acupressure Regimen

INTERVENTIONS:
Other: Acupuncture Regimen — Patients in the acupuncture and the acupressure group will receive a standardised treatment comprising 12 SEIRIN® press needles (with a sharp tip) at 7 acupuncture points (Du 26, He 9, Ren 17, bilateral LI 4, He 9, LV 3, Ma 36 and Pe 6). The point regimen is based on consensus process of national and international experts. All needling will be documented by the acupuncturist. Application time is supposed to be 84-96 hours. Modification, especially less points according to the patients reaction during treatment is allowed.
  Arms: Acupuncture Regimen
Other: Acupressure Regimen — Patients in the acupuncture and the acupressure group will receive a standardised treatment comprising 12 SEIRIN® press plasters (with a blunt knob instead a sharp needle) at 7 acupuncture points (Du 26, He 9, Ren 17, bilateral LI 4, He 9, LV 3, Ma 36 and Pe 6). The point regimen is based on consensus process of national and international experts. All needling will be documented by the acupuncturist. Application time is supposed to be 84-96 hours. Modification, especially less points according to the patients reaction during treatment is allowed.
  Arms: Acupressure Regimen

SUMMARY:
In the present study, the investigators want to evaluate if press needle acupuncture applied prior to surgery may contribute to the anaesthesiologic outcome. Acupuncture might improve fast-track anaesthesia in the PACU after general surgery.

DETAILED DESCRIPTION:
The use of complementary approaches, especially acupuncture, has gained momentum within the last decade. In this regard, it might be appropriate to develop a simply applicable (a) and effective (b) acupuncture regimen for the complementary support of fast-track anaesthesia. Regarding practicability (a), it might be of interest to reduce the amount of necessary acupuncture points. Trials have shown that single-point acupuncture is strong enough to cause relevant clinical effects (Fleckenstein et al., 2009; Lee and Fan, 2009). In addition, practicability means to reduce the amount of needling events; therefore the investigators suggest the use of press needles, making complete peri-anaesthetic availability possible. Regarding effectiveness (b), it has been reported that acupuncture at Governing Vessel 26 (Du-26) may be successful in shock resuscitation (Hsu et al., 2006). In combination with other points it has been evaluated in a Chinese study improving the vegetative state after operation of acute subdural hematoma (Zheng, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Scheduled for laparoscopic surgery of uterus, adnex or ovaries
* ASA-score ≤ 2
* Subjects with the ability to follow study instructions and likely to attend and complete all required visits
* Written informed consent of the subject

Exclusion Criteria:

General Exclusion Criteria:

* Subject without legal capacity who is unable to understand the nature, scope, significance and consequences of this clinical trial
* Simultaneously participation in another clinical trial or participation in any clinical trial involving administration of acupuncture within 30 days prior to clinical trial beginning
* Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the trial results, or may interfere with the subject's participation in this clinical trial
* Known or persistent abuse of medication, drugs or alcohol

Exclusion criteria regarding special restrictions for females:

* Current or planned pregnancy or nursing women
* Females of childbearing potential, who are not using and not willing to use medically reliable methods of contraception for the entire study duration (such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices) unless they are surgically sterilized / hysterectomized or there are any other criteria considered sufficiently reliable by the investigator in individual cases.

Indication specific exclusion criteria:

Subjects will not be included in the study if any of the following criteria applies:

* Surgery within the last three months
* Chronic pain > 3 month
* Continuous analgesic medication with opioids longer than 3 days
* Massive degenerative diseases
* Pre-treatment with acupuncture or trigger point injection within the last 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary objective is the assessment of the effects of permanent needle acupuncture at 12 acupuncture points for improving post anaesthetic recovery. | The time from extubation to "Ready for discharge" (in minutes) will followed for the duration in the recovery unit, an expected average of 1 hour
  Time from extubation to "Ready for discharge" (in minutes) from the PACU as assessed by the Aldrete score, the Post Anaesthetic Discharge Scoring System (PADSS) and our 'in-house' scoring system when comparing the acupuncture group and the standard treatment group.

SECONDARY OUTCOMES:
Preoperative Variables | 2 days, ends when anaesthesia starts
  Anxiety (STAI-Score)
Variables in PACU | Patients will be followed for the duration of their stay in the recovery unit, , an expected average of 1 hour
  Postoperative pain (pain intensity by VAS)
Postoperative variables | Patients will be followed for the duration of hospital stay follwing the recovery unit, an average of 2 days
  Postoperative pain (pain intensity by VAS)
Perioperative Variables | Patients will be followed for the duration of the surgical procedure, an expected average of 2 hours
  TCI effect concentrations
Perioperative Variables | Patients will be followed for the duration of the surgical procedure, an expected average of 2 hours
  Organizational time points (e.g. incision to closure time)

OTHER OUTCOMES:
Safety | 3 days
  Occurence of acupuncture side effects

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Irnich, PD Dr., Study Director — Department of Anaesthesiology, University of Munich
Locations (1):
- Department of Anaesthesiology, University of Munich, Germany., Munich, Bavaria, Germany

REFERENCES:
- [Background] Fleckenstein J, Sittl R, Averbeck B, Lang PM, Irnich D, Carr RW. Activation of axonal Kv7 channels in human peripheral nerve by flupirtine but not placebo - therapeutic potential for peripheral neuropathies: results of a randomised controlled trial. J Transl Med. 2013 Feb 8;11:34. doi: 10.1186/1479-5876-11-34. PMID 23394517
- [Derived] Fleckenstein J, Baeumler PI, Gurschler C, Weissenbacher T, Simang M, Annecke T, Geisenberger T, Irnich D. Acupuncture for post anaesthetic recovery and postoperative pain: study protocol for a randomised controlled trial. Trials. 2014 Jul 21;15:292. doi: 10.1186/1745-6215-15-292. PMID 25047046